CLINICAL TRIAL: NCT00205387
Title: Cardiac Elastography
Brief Title: Cardiac Elastography to Determine Strain and Strain Rates in the Heart
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: M-2004-1260
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2012-08-29 (Estimated); Status verified 2012-08

CONDITIONS: Heart Disease
Keywords: echocardiography; cardiac elastography; Normal volunteers
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: cardiac elastography and echocardiography — standard echocardiogram

SUMMARY:
Cardiac elastography is a new technique to analyze strain and strain rates in many organ systems, including the heart. In this study, cardiac elastography derived from the analysis of raw radiofrequency data obtained from a conventional clinical echocardiograph system will be compared to processed information that comes from the same echocardiograph system. The purpose of this study is to determine if cardiac elastography can accurately determine strain and strain rates as compared to more conventional means.

ELIGIBILITY:
Inclusion Criteria:

* Healthy normal volunteers between the ages of 18-70
* Patients scheduled for clinical echocardiogram between the ages of 18-70 who have known heart disease caused by myocardial infarction or cardiomyopathy

Exclusion Criteria:

* Patients less than 18 years old, or greater than 70 years old
* Patients who do not have adequate quality echocardiographic images.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy volunteers and patients with known heart disease caused by myocardial inarction or cardiomyopathy
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2005-11; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter S Rahko, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States